CLINICAL TRIAL: NCT04377074
Title: Parenting in a Pandemic: Parental Stress During the COVID-19 and Its Association With Depression and Anxiety
Brief Title: Parental Stress During the COVID-19 Pandemic and Its Association With Depression and Anxiety
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other); Oslo Metropolitan University (Other); University of Bergen (Other)
Responsible Party: Principal Investigator, Sverre Urnes Johnson, Associate Professor Sverre Urnes Johnson, University of Oslo
Other Study IDs: REK125510(3)
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Parental Stress; Depression; Anxiety
Keywords: COVID-19; Parental Stress; Social distancing; Quarantine; Isolation; Non-pharmacological interventions; Disease containment strategies; Depression; Anxiety; Worry
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to investigate the levels of parental stress across different demographic subgroups in the general parental population during the strict social distancing government-initiated non-pharmacological interventions (NPI's) related to the COVID-19 pandemic. The study also seeks to examine the predictors of parental stress rates related to these non-pharmacological interventions (NPI's). In addition, the research will investigate the association between parental stress associated and psychopathology symptoms (i.e., depression and generalized anxiety).

The aim of the project is to:

* Inform the policymakers, the general public, scientists, and health practitioners about the psychological associations of the COVID-19-related government-initiated measures on parental stress, with special focus on the school and kindergarten lockdowns.
* Provide a foundation for policymakers and health-care professionals to employ interventions that protect families against possibly increased psychological stressors.
* Help policymakers and healthcare professionals to better understand the association of demographic variables and other predictors on parental stress and parent-child dysfunction, which information necessary for evaluating the psychological impact of NPIs on parental stress and thus the framework under which decisions about school/kindergarten lockdowns are made.

DETAILED DESCRIPTION:
This study seeks to investigate the levels of parental stress across different demographic subgroups in the general parental population during the strict social distancing government-initiated non-pharmacological interventions (NPI's) related to the COVID-19 pandemic, including school and kindergarten lockdown. The study also seeks to examine the predictors of parental stress rates related to these non-pharmacological interventions (NPI's). In addition, the research will investigate the association between parental stress and psychopathology symptoms (i.e., depression and generalized anxiety) during the social distancing interventions.

The aim of the project is to:

* Inform the policymakers, the general public, scientists, and health practitioners about the psychological associations of the COVID-19-related government-initiated measures on parental stress, with special focus on the school and kindergarten lockdowns.
* Provide a foundation for policymakers and health-care professionals to employ interventions that protect families against possibly increased psychological stressors.
* Help policymakers and health-care professionals to better understand the association of demographic variables and other predictors on parental stress and parent-child dysfunction, information necessary in evaluating the psychological impact of social distancing measures on parental stress and thus the framework under which decisions about school/kindergarten lockdowns are made.

Hypothesis/Research Questions Hypothesis related to parental stress during the COVID-19 pandemic

1. H1: Gender (female), higher age, higher number of children, and having a pre-existing psychiatric diagnosis will be associated with more parental distress.

   a. We assume to find differences in parenting stress during the COVID-19 pandemic based on the existing literature on gender differences on parental behavior and distress (Scott & Alwin, 1989; Hildingsson & Thomas, 2013; Deater-Deckard & Scarr, 1996; McBride et al., 2002; Skari et al., 2002). The literature further suggests that higher age and higher number of children is associated with higher parental stress (Lavee et al., 1996; Östberg & Hagekull, 2000). Psychopathology symptoms, as reflected by having a pre-existing psychiatric diagnosis, is also found to be associated with parental stress (Pripp et al., 2010; Crugnola et al., 2016; Vismara et al., 2016; Leigh & Milgrom, 2008; Prino et al., 2016; Rollé et al., 2017).
2. H2: Worry and rumination in general, low self-efficacy, difficulty with working from home, burnout, low social support, and higher anger expression related to children are all associated with more parental distress, when age, number of children, gender and pre-existing psychiatric diagnosis are controlled for.

   a. Existing research literature have highlighted that perceived personal control is found to be directly related to parental stress (Guterman, 2009), and that women's levels of parental stress is related to parenting self-efficacy (Suzuki, 2010). Sepa and colleges (2004) also reported that lack of confidence/security were linked to parental stress. Reduced social support is also found to be associated with higher rates of parental stress (Östberg & Hagekull, 2000; Crnic et al., 1983; Suzuki, 2010; Koeske & Koeske, 1990; Sepa et al., 2004). Furthermore, anger expression is also found to be associated with parental stress in the existing research literature (Lam, 1999). We also hypothesize that burnout, worry and rumination in general and difficulty with working from home will be associated with higher parental stress, relations not previously explored in the existing literature.
3. H3: More parental distress will be associated with more depressive symptoms and anxiety symptoms, when gender, pre-existing psychiatric diagnosis, age and number of children are controlled for.

   1. Previous studies have found that parents with psychological problems, such as depression and generalized anxiety disorder, are at greater risk for parenting stress, and that parental stress may result in depression and anxiety (Pripp et al., 2010; Crugnola et al., 2016; Vismara et al., 2016; Leigh & Milgrom, 2008; Prino et al., 2016; Rollé et al., 2017).

Exploratory: Additionally, we will investigate the differences in levels of parental distress across different demographic subgroups in the sample.

Participants were asked to fill out a set of validated questionnaires including demographic variables, psychological symptoms, situational factors related to the consequences of the COVID-19 virus, personality-trait and, and worry, in a random order. Some questionnaires are given as a whole, whereas other questions include theoretically driven selections of items from validated questionnaires, based on a panel of clinical experts, with the goal of avoiding topological overlap. This study is part of a 'The Norwegian COVID-19, Mental Health and Adherence Project' involving multiple studies. In order to not overwhelm and burden the participants with long questionnaire, and due to the mentioned empirical concerns of topological overlap (i.e., overlap in item content) between similar items (for network analysis purposes), in some scales involving large item-content overlap, single items were chosen in a theory-driven manner by three independent clinical psychologists and clinical specialists in adult psychopathology.

Data collection started during the time-period with the strictest and equal number of government-initiated non-pharmacological interventions (NPI's) in Norway, and data collection was stopped once these NPI's were modified or new information about NPI's were added. The data include one directly identifiable variable (contact information) for participants in accordance to the General Data Protection Regulation (GDPR) law in EU, which is to give the participants the opportunity to have their data deleted upon request. Data are thus kept on a safe server belonging to the University of Oslo and will be accessed first following de-identification. Stopping rule for data collection: Stopping rule: 1) At once if government-initiated NPI's are modified or novel information are given about NPIs (to control for cognitive variables) and/ or 2) once we reach enough participants given the power analysis.

Measures: PHQ-9; GAD-7; parental stress; demographic variables (gender; age; civil status; employment status; education level; number of children in household); situational variables (difficulty to work from home; burnout; anger expression related to children; social support; worried or ruminated on problems); person-trait variables (self-efficacy ("I can always manage to solve difficult problems if I try hard enough) and whether one has a psychiatric diagnosis or not. The self-efficacy item is chosen from The General Self-Efficacy Scale (Tambs & Røysamb, 2014). The parental stress subscale is based on three items from the Danish Parental Stress Scale (Potoppidan et al., 2018).

The outcome variables are Parental Stress, consisting of a total score of parental stress based on items from the Danish parental stress scale; PHQ-9; GAD-7. The other variables are predictors of these three outcome variables. For the parental stress regression analyses we will include the following variables: age, gender, number of children in household, psychiatric diagnosis, difficulty to work from home, worry and rumination; anger expression related to children, social support and self-efficacy. The other two multiple regression analysis will investigate whether parental stress is associated with depression and anxiety symptoms while controlling for the following variables: gender, age, number of children in household and psychiatric diagnosis.

Inference criteria:

Given the large sample size, the investigators pre-defined our significance level:

p< 0.01 to determine significant.

Sample size estimation:

The mentioned 'Norwegian COVID-19, Mental Health and Adherence Project' involves multiple studies, where some involve a Complex Systems (Network analysis) approach. These mutlivariate analyses require large samples and power analysis was conducted accordingly. Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants be at the very least three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. Thus, with the more conservative estimates by Roscoe, an optimal sample size for the specific study on parents included more than 2530 individuals. According to the stopping rule mentioned above, due to the importance of keeping the NPI variable constant, we would stop data collection even if we did not obtain our target N. Fortunately, sufficient sample was reached during a period with identical NPIs across the country.

Statistical analyses:

Three multiple regression analysis will be conducted; one with parental stress; the second and third with PHQ-9 and GAD total scores as dependent variables. Specific predictors for these three multiple regression analyses are listed above (hypothesis section). Multicollinarity and other assumptions will be checked; if the multicollinearity is violated (if VIF > 5 and Tolerance > 0.2; Hocking, 2003); O'Brian, 2007).

Note that this the project outline, study plan and analysis was registered upon application to the Regional Committees for Medical and Health Research Ethics (REC) and Norwegian Centre for Research Data 10 days prior data collection, two committees which evaluate the rational for data collection and hypotheses as well as evaluate the ethical aspects of the study before allowing the data to be collected. The study is registered on clinicaltrials.gov after completed data collection, although this registration is prior to any analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

- Eligible participants are all parents (over 18 years) living with one or more child under 18 years, and/or a child over 18 with special needs (i.e. physical disabilities). All participants are currently living in Norway and thus experiencing identical NPIs, and who had provided digital consent to partake in the study.

How the participants were reached:

Given the time-sensitivity of the project and the strict and time-consuming process of getting approval to access registry data, the investigators did not apply for access to registry data (e.g., address, phone or e-mails of the general population), as such data access is highly strict and regulated in Norway and the time-frame of such an application could have encompassed variation in an important variable we wished to hold constant (namely identical NPIs (non-pharmacological interventions) employed over the time-frame of data collection). Thus, the investigators did not apply for registry data, reached out the population through the means elaborated below. The investigators reached out to the general Norwegian population systematically in the following six ways, with the goal of providing the entire adult population an equal opportunity to be exposed to the survey:

1. Through broadcasting on the main national news channel of Norway which had nearly 1.1 million viewers at the time of broadcast.
2. Using Facebook Business Advertisement where we exposed all adult Norwegian Facebook users (3.6 million; 85% of the Norwegian adult population) with an equal opportunity of being exposed to the survey in a random manner. Our survey reached a random selection of nearly 180 000 of the adult population.
3. Broadcasting the survey on national and region radio stations across the country
4. Broadcasting about the survey on local radio stations across the country
5. Using national newspaper to reach out to participants about the survey
6. Using regional and local newspapers to reach out to participants across all regions and counties in Norway.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Biological Sex and self-representation of gender are measured. All participants are welcome to partake in the study.
Study Population: The general population of parents (Age >= 18) from all regions (i.e., counties) of Norway, having equal opportunity and the probability of partaking in the study.
Sampling Method: Probability Sample
Enrollment: 2880 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Measure of parental stress | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  Three items from the Danish Parental Stress Scale (PSS) was selected, which intends to be a short measure of perceived stress resulting from being a parent (Pontoppidan et al., 2018). The scale consists of nine items measuring parental stress where each is measured on a five-point Likert scale (1-5), with the scores ranging from 3 to 15. Higher scores indicate higher parental stress. The following three were chosen in this large-scale investigation: 1) I feel overwhelmed by the responsibility of being a parent. 2) The major source of stress in my life is my child(ren), and 3) It is difficult to balance different responsibilities because of my child(ren) (Pontoppidan et al., 2018).
Patient Health Questionnaire 9 | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27. Higher scores indicate greater depression severity, and scores above 10 are considered as the cut-off that indicating that the patient is within the depressive area.
Generalized Anxiety Disorder 7 | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21. Higher scores indicate greater anxiety severity, and scores that are above the cutoff of 10 are considered to be in the clinical range (Spitzer et al., 2006). Specific cut-off for Norwegian samples have been found yielding a cut-off of 8 and above for high sensitivity and specificity (Johnson, Ulvenes, Øktedalen & Hoffart, 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Sinkerud Johnson, PhD, Principal Investigator — Oslo Metropolitan University; Nora Paulsen Skjerdingstad, Principal Investigator — University of Bergen; Omid Ebrahimi, Principal Investigator — University of Oslo & Modum Bad; Asle Hoffart, PhD, Principal Investigator — Modum Bad & University of Oslo; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo & Modum Bad
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No